CLINICAL TRIAL: NCT00000132
Title: Early Manifest Glaucoma Trial (EMGT)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Eye Institute (NEI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: NEI-31
Record Dates: First submitted 1999-09-23; First posted 1999-09-24 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-10

CONDITIONS: Open-Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Betaxolol

INTERVENTIONS:
Drug: Betaxolol
Procedure: Argon Laser Trabeculoplasty

SUMMARY:
The primary purpose is to compare the effect of immediate therapy to lower the intraocular pressure (IOP) versus late or no treatment on the progression of newly detected open-angle glaucoma, as measured by increasing visual field loss and/or optic disc changes.

The secondary purposes are to determine the extent of IOP reduction attained by treatment, to explore factors that may influence glaucoma progression, and to describe the natural history of newly detected glaucoma.

DETAILED DESCRIPTION:
Glaucoma is a common disease in older adults. All present treatment aims at reduction of the intraocular pressure, but indications for therapy are not well defined. Furthermore, it is unclear whether intraocular pressure influences the natural history of glaucoma. Against this background, the primary aim of the study is of central importance to patients with manifest and suspect glaucoma.

Glaucoma has few subjective symptoms during a long period early in the disease, but damage is irreversible once it occurs. Early diagnosis and rapid detection of progression are of paramount importance in limiting this damage, whether through pressure reduction or in some other way. The effectiveness, if any, of lowering the intraocular pressure in glaucoma requires evaluation by controlled treatment trials.

The Early Manifest Glaucoma Trial (EMGT) is the first large, controlled, randomized clinical trial to evaluate the effect of lowering the intraocular pressure on the progression of newly detected, open-angle glaucoma. This study will compare glaucoma progression in initially treated versus untreated patients with newly detected open-angle glaucoma and will allow quantification of the effect of immediate IOP-lowering treatment on progression during the followup period.

The EMGT is a collaborative effort that involves a Clinical Center at the Department of Ophthalmology of Malmo University Hospital at the University of Lund, Sweden, and its Satellite Center in Helsingborg, Sweden; an independent Data Center at the Department of Preventive Medicine, University Medical Center at Stony Brook, New York; and a Disc Photography Reading Center at the Department of Ophthalmology in Lund at the University of Lund. The study was initiated with support from the Swedish Medical Research Council.

Recruitment for the study has been completed. The 255 patients were identified by an extensive, population-based screening of successive age cohorts as well as by clinical referral. The diagnosis was confirmed through Humphrey perimetry at two postscreening visits to the Clinical Center or Satellite Center. Eligible patients who agreed to participate had two additional visits for collection of baseline data. They were randomized to treatment with the beta blocker Betaxolol and argon laser trabeculoplasty (treated group) or to no initial treatment (control group) with close followup of both groups.

Patients are followed for a minimum of 4 years to assess the development of glaucoma progression. They are seen every 3 months to collect visual field, IOP, and other data. Disc photographs are taken every 6 months. Technicians and disc photograph graders are masked regarding treatment assignment. Additional followup visits are held to confirm visual field progression and IOP elevation (>25 mm Hg in treated group, >35 mm Hg in control group). Patients in the treated group receive Xalantan whenever IOP exceeds 25 mm Hg at more than one visit; patients in the control group will receive Xalantan whenever IOP reaches 35 mm Hg or higher during the trial. If IOP remains high, individualized treatment is given. All patients continue to be followed to monitor the development of end points and will be analyzed in their originally assigned groups.

The study outcome is glaucoma progression, which is based on specific criteria derived from analyses of Humphrey visual fields and masked evaluations of disc photographs. The perimetric outcome is defined as statistically significant deterioration (p < 0.05) of the same three or more test points in Pattern Deviation Change Probability Maps in three consecutive C30-2 Humphrey fields. Optic disc progression is determined by the following:

* The presence of definite change (detected by comparison of followup photographs with baseline) by flicker chronoscopy in two followup photographs from the same visit, with independent confirmation by side-by-side gradings.
* Final confirmation of change toward progression, by flicker chronoscopy and by side-by-side gradings, at a different followup visit.

ELIGIBILITY:
Men and women between ages 50 and 80 years who have newly detected and untreated chronic open-angle glaucoma with repeatable visual field defects by Humphrey perimetry are eligible for inclusion.

Exclusion criteria include the following: advanced visual field loss (MD less than or equal to 16 dB) or threat to fixation; mean IOP > 30 mm Hg or any IOP > 35 mm Hg in at least one eye; VA < 0.5 in either eye; or any conditions precluding reliable fields or photos, use of study treatment, or 4-year followup.

Ages: 50 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 1992-10

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Department of Ophthalmology, Helsingborg Hospital, Helsingborg
  - Department of Ophthalmology, Malmo University Hospital, University of Lund, Malmo

REFERENCES:
- [Derived] Rolim-de-Moura CR, Paranhos A Jr, Loutfi M, Burton D, Wormald R, Evans JR. Laser trabeculoplasty for open-angle glaucoma and ocular hypertension. Cochrane Database Syst Rev. 2022 Aug 9;8(8):CD003919. doi: 10.1002/14651858.CD003919.pub3. PMID 35943114
- [Derived] Heijl A, Peters D, Leske MC, Bengtsson B. Effects of argon laser trabeculoplasty in the Early Manifest Glaucoma Trial. Am J Ophthalmol. 2011 Nov;152(5):842-8. doi: 10.1016/j.ajo.2011.04.036. Epub 2011 Aug 16. PMID 21843876